CLINICAL TRIAL: NCT06321718
Title: Comparison Between Pericapsular Nerve Group (PENG) Block With Lateral Femoral Cutaneous Nerve Block and Supra Inguinal Fascia Iliaca Compartment Block (S FICB) for Traumatic Hip Fixation Surgeries: a Randomized Controlled Trial
Brief Title: Pericapsular Nerve Group Block vs Supra Inguinal Fascia Iliaca Compartment Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Abd El-Khalek Mohammed Glala, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04-2023-200629
Record Dates: First submitted 2024-02-21; First posted 2024-03-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: 96 Patients will be enrolled. Choice of type of anesthesia will be established according to every individual patient, but spinal anesthesia will be preferred over general anesthesia. The block will be administered under supervision of the supervisor senior staff before induction of anesthesia. 2 groups well be assessed
  1. Group (A) will receive PENG + LFCN block
  2. The second group (B): S-FICB
Who Masked: Participant
Masking Description: Through website computer program randomization program to distribute cases into two groups using their order number
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Group (A) (Experimental): will receive PENG + LFCN block
- 2. group (B) (Experimental): will receive S-FICB

INTERVENTIONS:
Procedure: PENG + LFCN block versus S-FICB — 1. Group (A) will receive PENG + LFCN block:

SUMMARY:
This study aims to assess the efficacy of PENG block performed with LFCN block in controlling postoperative pain and promoting motor function recovery and to compare its effectiveness with S-FICB.

DETAILED DESCRIPTION:
96 Patients will be assessed thoroughly for history (to exclude previous medical history, previous anesthesia, with/without perioperative complications, smoking status, cardiorespiratory disorders or bleeding disorders), examination (for the full primary and secondary trauma survey to exclude any coexisting trauma that threatens patient life, laboratory (for CBC, bleeding tendencies, serology, kidney dysfunction and availability of blood transfusion) and radiological (for cardiac assessment, and exclusion of other trauma). ASA score then to be determined. Full monitoring of the patient will be recorded, basically, HR, ECG, SpO2, NIBP, EtCO2, temperature. Peripheral vein cannula will be secured and the fluids will be infused as 10- 15ml/kg before induction of anesthesia. Choice of type of anesthesia will be established according to every individual patient, but spinal anesthesia will be preferred over general anesthesia. The block will be administered under supervision of the supervisor senior staff before induction of anesthesia. Type of the block will be randomly assigned into two groups according to website computer program randomization program to distribute cases into two groups using their order number:

1. Group (A) will receive PENG + LFCN block: The low-frequency curvilinear probe (3-5 MHz) of ultrasound (GE Logiq e, GE Health care, USA) will be placed in a transverse plane over the anterior inferior iliac spine (AIIS) and aligned with the pubic ramus by rotating the probe counterclockwise to obtain a hyper-echoic bright line, which is the iliopubic eminence (IPE). In this view, the iliopsoas muscle and psoas tendon, the femoral artery, and pectineus muscle can be observed. Using the in-plane injection technique, a 22G, 80 mm insulated block needle was inserted in a lateral-to-medial direction, and the tip will then be placed between the psoas tendon anteriorly and the pubic ramus posteriorly. After no blood was drawn back, the LA (20 ml, 0.25% bupivacaine) will be injected to get an image of the psoas tendon uplifted. After the PENG block is performed, a high-frequency linear probe (6-12 MHz) will be placed on the inguinal ligament to get a short-axial view of femoral artery, then the probe is moved laterally to identify the sartorius muscle, the tail of the probe will be positioned toward the anterior superior iliac spine to observe the LFCN covered by fascia between sartorius and tensor fascia lata. After no blood can be withdrawn back, the LA (10 ml, 0.25% bupivacaine) will be injected following negative aspiration
2. The second group (B): S-FICB: A high-frequency linear probe (6-12 MHz) of ultrasound (GE Logiq e, GE Healthcare, USA) will be used. The probe is placed adjacent to the inguinal ligament with its long axis parallel to the ligament. After the femoral artery and the femoral nerve will be observed, the probe will be moved laterally to identify the sartorius muscle and placing it at the center of the screen. Then the probe will be moved cephalically to the anterior superior iliac spine (ASIS) until the image of the sartorius muscle will disappear, and the medial side of ASIS was identifed as the iliacus muscle. Next, by rotating the medial end of the ultrasound probe toward the umbilicus, the ASIS, iliac bone, and abdominal muscles will be observed on the screen. Using the in-plane technique, a 22G, 80 mm insulated block needle will be inserted in a lateral-to-medial direction. When the needle tip will penetrate below the fascia iliacus, the LA (40 ml, 0.25% bupivacaine) will be injected following negative aspiration to obtain an image showing the LA spread between the iliacus muscle and the fascia iliacus.

ELIGIBILITY:
Inclusion Criteria:

1. All hip trauma patients ≥ 18 years' old
2. ASA class I, II, and III
3. Solitary hip fracture

Exclusion Criteria:

1. Neurological disturbance either baseline or traumatic brain injury
2. Contraindications for regional anesthesia as bleeding disorders, infection at site of injection, or hypersensitivity to the used local anesthetics.
3. Patient refusal.
4. Massive poly trauma.
5. Uncooperative patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
recording time for "return of full muscle power" | at hour 0, 2 hours, 4 hours, 6 hours, 12 hours after procedure
  duration between the end of surgery and the first time the patient was able to move his operated leg. The full power return will be defined as pre-operative muscle power according to manual muscle testing scale (MRC)/ Muscle Power Scale as following: Score Description 0 No contraction
  1. Flicker or trace of contraction
  2. Active movement, with gravity eliminated
  3. Active movement against gravity
  4. Active movement against gravity and resistance
  5. Normal power

SECONDARY OUTCOMES:
• The degree of hip flexion on the operative side | at 6 hours, 24 hours, and 48 hours.
  • The degree of hip flexion on the operative side ( full range, mild restriction, major restriction, or completely no movement)
• Static and dynamic pain scores. | at 6 hours, 24 hours, and 48 hours.
  A person rates their pain on a scale of 0 to 10 or 0 to 5. Zero means "no pain," and 5 or 10 means "the worst possible pain." These pain intensity levels may be assessed upon initial treatment, or periodically after treatment
postoperative nausea and vomiting (PONV) scale | at 48 hours.
  no nausea (0), mild nausea with no treatment need (1), moderate nausea and vomiting with need to treatment (2), severe nausea and vomiting even with treatment (3)
• The number of rescue analgesia | 24 hours
  Times that he needs analgesic 30 mg ketorolac

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, faculty of medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR